CLINICAL TRIAL: NCT04943367
Title: Efficacy of TEAS On Prevention of Rocuronium Injection Pain
Brief Title: Effect of TEAS on Rocuronium Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Rocuronium injection pain
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Injection Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP TEAS (Active Comparator): Patients will receive TEAS bilaterally at two acupoints: Hegu (L14) and Neiguan (PC6).
  Interventions: Device: TEAS
- Control Sham Group (Placebo Comparator): Patients in the sham group will be undergoing electrode attachment on the target acupoints without electronic stimulation.
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS — Transcutaneous electrical acupuncture stimulation

SUMMARY:
Pain from the injection of rocuronium is a common side effect during anesthetic practice, occurring in 50%-80% of patients. Several methods have been used to reduce this pain. This prospective, randomized study was designed to determine the efficacy of transcutaneous electrical acupuncture point stimulation in reducing the rocuronium injection pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year aged
* ASA I-III
* Who was to undergo various elective operations.

Exclusion Criteria:

* Cardiovascular surgery
* Patients with pacemakers
* Patients requiring rapid sequential induction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Pain with rocuronium injection | 5 minutes
  pain will be graded as no pain; mild pain; moderate pain; severe pain following administration of a priming dose of rocuronium

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)